CLINICAL TRIAL: NCT04067804
Title: Cultivating Healing by Implementing Restorative Practices for Youth
Brief Title: Implementing Restorative Practices for Youth
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the project could no longer be implemented effectively and with fidelity
Sponsor: Pacific Institute for Research and Evaluation (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency); University of California, San Diego (Other); Restorative Solutions, Inc. (Unknown); Western Implementation Research and Evaluation (Unknown)
Responsible Party: Principal Investigator, Cathleen Willging, Senior Research Scientist II and Center Director, Pacific Institute for Research and Evaluation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 08740101; 2016-CK-BX-0008 (Other Grant/Funding Number: National Institute of Justicie)
Record Dates: First submitted 2018-05-15; First posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Discipline Practices
Keywords: Implementation Research; School-based research; Restorative Practices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Standard school disciplinary practices.
- Dynamic Adaptation Process (Experimental): Using the Dynamic Adaptation Process, specialist coordinators will convene and lead Implementation Resource Teams (IRTs). With the assistance of expert trainers and coaches, the coordinator-led IRTs will then engage in an iterative process of assessment and planning to build school capacity and implement restorative practices to reduce adverse student outcomes related to discipline.
  Interventions: Behavioral: Dynamic Adaptation Process

INTERVENTIONS:
Behavioral: Dynamic Adaptation Process — The Dynamic Adaptation Process draws from implementation science frameworks and methods, including the Exploration, Preparation, Implementation, and Sustainment model, to organize planning and implementation activities. The Dynamic Adaptation Process is a structured methodology designed to integrate new interventions within complex systems, such as schools.
  Arms: Dynamic Adaptation Process

SUMMARY:
1.1 Project Goals and Objectives: The goals for this project are to: (1) Engage school district stakeholders in a Southwestern U.S. state in a structured planning process for incorporating tailored restorative practices within culturally and economically diverse middle schools to reduce adverse student outcomes related to discipline; (2) Produce scientific evidence regarding the effectiveness and the costs/benefits of restorative practices implemented in these middle schools using a stratified cluster randomized design and mixed methods; and (3) Build capacity within schools to implement and evaluate restorative practices with fidelity after implementation support has ended, and to facilitate a cascade of practices districtwide. The project consists of four phases based on the Exploration, Preparation, Implementation, and Sustainment (EPIS) model.

DETAILED DESCRIPTION:
Statement of the problem: Zero-tolerance policies, emphasizing rigid responses to infractions, including removal of students from school and referrals to juvenile justice systems, have prevailed nationwide. Such policies disproportionately affect minority/disadvantaged students by severely disciplining them for minimal infractions, imperiling their academic performance and graduation, and potentially leading to detention or incarceration. In contrast, restorative justice practices elicit understanding of the perspectives of those involved in conflict and rule violations, addressing the effect of offenses, and remedying the damage, thus opening up healing opportunities and keeping students in the classroom. Yet, little research exists regarding their effectiveness in reducing negative student outcomes and developing positive school climates. Our knowledge of factors associated with successful implementation and fidelity, and adaptations at the district, school, staff, and student levels to promote their sustained use is also inadequate.

Partnerships: This project addresses these gaps by developing a Community-Academic Partnership (CAP) to implement and evaluate a large-scale restorative practice initiative for middle schools. Our CAP involves a Southwestern U.S. state school district that wishes to remain anonymous, other key community entities, and academic researchers.

Research design/methods: The project will: (1) Engage school district stakeholders in a structured planning process for incorporating tailored restorative practices within culturally and economically diverse middle schools to reduce adverse student outcomes related to discipline; (2) Produce scientific evidence regarding the effectiveness and the costs/benefits of restorative practices implemented in these middle schools using a stratified cluster randomized design and mixed methods; and (3) Build capacity within schools to implement and evaluate restorative practices with fidelity after implementation support has ended, and to facilitate cascade of practices districtwide. A combination of qualitative methods (interviews, focus groups, and document review) and quantitative methods (surveys and administrative data review) will be used to evaluate and track implementation success and outcomes.

Analysis: Procedures include iterative qualitative data coding, descriptive statistical analysis, multilevel modeling, and cost/benefits analysis.

Products, reports, and archiving: This project will advance a set of strategies to enhance child wellbeing. The CAP will disseminate these strategies and accompanying evaluation methods via national/state conferences, districtwide reports, peer-reviewed publications, and open access mediums.

ELIGIBILITY:
Inclusion Criteria:

* Middle school in the school district of study (School district wishes to remain anonymous)

Exclusion Criteria:

* A school that is not a middle school in the school district of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Student Disciplinary Actions | 1 year. Change from baseline through study completion, an average of 48 months
  Outcomes include total number of (1) detentions, (2) in-school suspensions, (3) out-of-school suspensions, (4) expulsions, and (5) referrals to juvenile justice.
Bullying | 24 months. Change from baseline, through study completion, an average of 48 months
  Measured by the state's Youth Risk Behavior Surveillance System Survey, outcomes will include student reports of bullying in the past 12 months.
School Safety | 24 months. Change from baseline, through study completion, an average of 48 months
  Measured by the state's Youth Risk Behavior Surveillance System Survey, outcomes will include student reports of missing school in the past 30 days due to fears about their safety.
Teacher Support | 24 months. Change from baseline, through study completion, an average of 48 months
  Measured by the state's Youth Risk Behavior Surveillance System Survey, outcomes will include student reports of a teacher or other adult at their school that makes them feel supported.

SECONDARY OUTCOMES:
Implementation Progress | 1 year. Change from baseline through study completion, an average of 48 months
  Progress will be measured using a modified Stages of Implementation Completion (SIC) checklist. The SIC is an eight-stage measure that assesses progress of implementation using activity completion dates and duration of activities.
Implementation Fidelity | 30 days. Change from baseline through study completion, an average of 48 months
  The specialist coordinators will conduct monthly fidelity ratings using a standardized checklist and provide data to their Implementation Resource Teams. A school staff web-survey across all 12 middle schools will also examine how frequently staff participate in the five primary restorative practice techniques and the level of perceived school support for these practices.
Cost/Benefit Analysis | Change from baseline through study completion, an average of 60 months
  Adhering to 2016 National Academy of Sciences guidelines, the intervention Cost/Benefit Analysis will focus on existing return on investment from both societal and government perspectives.

CONTACTS AND LOCATIONS:
Overall Officials: Cathleen Willging, Ph.D., Principal Investigator — Pacific Institute for Research and Evaluation
Locations (1):
- Pacific Institute for Research and Evaluation, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No